CLINICAL TRIAL: NCT00473954
Title: A Phase 1, Open-Label, Dose Escalation Study of the Safety and Preliminary Efficacy of EGEN-001 in Combination With Carboplatin and Docetaxel in Women With Recurrent, Platinum-Sensitive, Epithelial Ovarian Cancer
Brief Title: Safety and Efficacy of EGEN-001 Combined With Carboplatin and Docetaxel in Recurrent, Platinum-Sensitive, Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EGEN, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGEN-001-201
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — GEN-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EGEN-001 (Experimental)
  Interventions: Genetic: EGEN-001 (phIL-12-005/PPC)

INTERVENTIONS:
Genetic: EGEN-001 (phIL-12-005/PPC) — In stage 1, patients will receive standard doses of IV carboplatin and docetaxel for 2 treatment cycles with a 3 week interval. Patients will also receive 4 IP infusions of EGEN-001 at 12mg/m2 EGEN-001, 18mg/m2, or 24mg/m2, 10-11 days apart.
  Stage 2 of the study will involve cycle escalation at the highest EGEN-001 dose identified from Stage 1. All patients will receive up to 8 doses of EGEN-001, 10-11 days apart plus up to 4 IV carboplatin and docetaxel cycles with 3 week intervals. After receiving the assigned number of treatments of EGEN-001, carboplatin, and docetaxel, patients may continue to receive up to 4 additional infusions of EGEN-001 and 2 IV carboplatin and docetaxel cycles with 3 week intervals.

SUMMARY:
Ovarian cancer may be caused by a build-up of genetic defects, or damaged genes within the body's cells. When genes are damaged, the body may be unable to produce a group of proteins, called cytokines, used by the immune system to fight cancer and some infections. The investigational gene transfer agent EGEN-001 contains the human gene for the cytokine interleukin-12 (IL-12) in a special carrier system designed to enter the cells and help the body to produce cytokines. Therefore, the purpose of the EGEN-001 therapy is to attempt to enhance the body's natural ability to recognize and fight cancer cells. Funding Source - FDA OOPD

DETAILED DESCRIPTION:
This study has two purposes:

* To determine what different strengths and number of doses of EGEN-001, administered directly into the peritoneal cavity, can be given safely in combination with standard intravenous chemotherapy for ovarian cancer
* To evaluate the anti-cancer activity of EGEN-001 when combined with standard chemotherapy; biological markers of EGEN-001 activity will be collected and ovarian cancer burden will be evaluated per standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Be female and at least 18 years of age (or minimum legal age and competency to provide voluntary written informed consent for study participation);
* Histologically/cytologically confirmed epithelial ovarian cancer that meets one of the following criteria:
* measurable disease by computed tomography (CT) scan or
* malignant ascites, or
* Serum CA-125 levels; or
* Clinically evaluable recurrent disease by other criteria.
* Relapsed, platinum-sensitive, ovarian cancer after induction chemotherapy (at least 6 months since last exposure to platinum based therapy).
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0, 1 or 2;
* Recovered from prior chemotherapy, having adequate bone marrow function:
* Adequate renal function;
* Adequate liver function;
* If of childbearing potential, have a negative pregnancy test and agree to follow an acceptable method of birth control;
* Agree to be compliant with the study's requirements;
* Understand and sign a written Informed Consent prior to the performance of any study-related procedures.

Exclusion Criteria:

* Ovarian cancer other than documented epithelial cancer;
* Intra-abdominal disease > 5 cm in diameter;
* Any serious, uncontrolled, intercurrent medical illness or disorder including, but not limited to:

  * Autoimmune disorders
  * Cardiac Disorders
  * Diabetes
  * Intrahepatic disease/cancer as documented by CT-scan
* An active infection within 4 weeks of study entry;
* Any condition/anomaly that would interfere with the appropriate placement of the IP catheter for study drug administration
* Prior treatment with whole abdominal irradiation;
* Currently receiving or have received any investigational agents within 28 days of study entry;
* Received prior chemotherapy for ovarian cancer administered by the IP route;
* Received any chemotherapy between completion of primary chemotherapy for ovarian cancer and study entry (e.g. consolidation therapy);
* Receipt of immunotherapy and/or any medications with the potential to affect the activity of EGEN 001;
* Known history of HIV infection, hepatitis B, or hepatitis C;
* Known hypersensitivity to any of the components of carboplatin or docetaxel;
* Life expectancy of less than 3 months;
* Known, current, recreational drug or alcohol abuse;
* Breast feeding an infant;
* Psychiatric illness/social situations which would limit compliance with study requirements;
* Any other known condition which in the Investigator's opinion would make the patient a poor candidate for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Determine the MTD and treatment-related toxicities of intra-peritoneal (IP) infusion of EGEN-001 in combination with carboplatin and docetaxel for recurrent, platinum-sensitive, ovarian cancer. | 12-14 months

SECONDARY OUTCOMES:
Examine the optimal EGEN-001 treatment regimen in combination with carboplatin and docetaxel in recurrent, platinum-sensitive ovarian cancer, and assess EGEN-001's impact on tumor, CA-125, and activity markers of biological activity. | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D. Alvarez, MD, Principal Investigator — Division of Gynecologic Oncology at University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Oncology Specialties, PC, Huntsville, Alabama
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas